CLINICAL TRIAL: NCT05454098
Title: A Food Effect Phase I Study of the Clifutinib in Healthy Subjects
Brief Title: Clifutinib Food Effect Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HEC73543-AML-103
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2022-07

CONDITIONS: Acute Myeloid Leukemia in Children

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fed states in healthy subjects (Experimental): A single 40mg dose of Clifutinib administered in a fed state.
  Interventions: Drug: Clifutinib with fed state
- Fasted states in healthy subjects (Experimental): A single 40mg dose of Clifutinib administered in a Fasted state.
  Interventions: Drug: Clifutinib with fasted state

INTERVENTIONS:
Drug: Clifutinib with fed state — 40 mg Clifutinib with food
  Arms: Fed states in healthy subjects
Drug: Clifutinib with fasted state — 40 mg Clifutinib without food
  Arms: Fasted states in healthy subjects

SUMMARY:
The purpose of this study is to evaluate to determine the effect of food on the PK of a single dose of 40 mg Clifutinib in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects (male or female), age greater than or equal to 18 years and less than or equal to 45 years;
* Weight ≥50 kg (≥45 kg for female), and have a body mass index (BMI) between 18 and 28 (including 18 and 28) at screening;
* Physical examination, clinical laboratory examination and other related examinations are normal or acceptable deviations that are judged to be not clinically significant by the investigator;
* Male or female subjects with child-bearing potential must agree to use effective contraception during the study and within 6 months after the administration of the last dose, and sperm donation is not allowed for male subjects during the study; female subjects must be non-pregnant and non-lactating；
* Volunteer to participate in this study, understand the study procedures and sign the informed consent prior to any study specific procedures, good compliance and willing to follow study procedures.

Exclusion Criteria:

* Have a history of or current cardiovascular, respiratory, hematological, hepatic, renal, gastrointestinal, endocrine, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs;
* Unable to tolerate standard meals;
* Prolonged QT interval corrected for heart rate using Fridericia's formula (QTcF) >470 ms (female >480 ms), or history of long QT syndrome；
* Have received live vaccine(s) within 3 months prior to screening;
* Have used over-the-counter or prescription medication , including herbal medications, within 14 days prior to dosing and during the study;
* Have known allergy to any drug or food;
* Smoking more than 5 cigarettes per day (or equivalent in tobacco or nicotine products) within 3 months prior to screening, or unwilling to abide by smoking restrictions during the study;
* Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody ,human immunodeficiency virus (HIV) antibody or Treponema pallidum antibody;
* Known history of drug abuse

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Cmax | 4 weeks
  Pharmacokinetics parameters in fasting state and fed state
AUC0-∞ | 4 weeks
  Pharmacokinetics parameters in fasting state and fed state

SECONDARY OUTCOMES:
Adverse Events | Through study completion, an average of 4 weeks
  Safety and tolerability measure by number of subjects who experience adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Derived] Wang D, Wu M, Li X, Jiang Y, Liu B, Zhang Y, Deng L, Ding Y. A phase I study of HEC73543, an oral FLT3 inhibitor: the effect of food on pharmacokinetics after oral dosing in healthy Chinese volunteers. Front Pharmacol. 2025 Oct 8;16:1636504. doi: 10.3389/fphar.2025.1636504. eCollection 2025. PMID 41069609